CLINICAL TRIAL: NCT00909519
Title: A Phase 1, Single-Center, Randomized, Parallel-group, Placebo- and Naproxen- Controlled, Double-blind Study to Evaluate the Effect of Naproxcinod 750 mg Bid Administered for 8 Days on the Renal Hemodynamics, Natriuretic and Renin Responses to a Single Bolus IV Dose of Furosemide 40 mg in Male Healthy Normotensive Volunteers
Brief Title: Effect of Repeated Dosing of Naproxcinod on Renal Hemodynamic and on Sodium Balance in Healthy Volunteers Before and After a Single Dose of Furosemide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NicOx (Industry)
Responsible Party: NicOx, NicOx
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: HCT3012-X-113
Record Dates: First submitted 2009-05-27; First posted 2009-05-28 (Estimated); Last update posted 2011-06-17 (Estimated); Status verified 2011-06

CONDITIONS: Renal Hemodynamics
MeSH Terms: interventions — naproxen-n-butyl nitrate; Naproxen; Furosemide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- naproxen (Active Comparator)
  Interventions: Drug: Naproxen
- naproxcinod (Experimental)
  Interventions: Drug: naproxcinod; Drug: furosemide
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: naproxcinod — naproxcinod 750 mg bid
  Arms: naproxcinod
Drug: Naproxen — Naproxen 500 mg bid
  Arms: naproxen
Drug: placebo — placebo
  Arms: placebo
Drug: furosemide — furosemide
  Arms: naproxcinod

SUMMARY:
This phase 1 study is an 8-day treatment period, randomized, controlled, double-blind, 3 parallel-groups, monocentric study. The primary objective is to evaluate the effect of naproxcinod on the renal function when co-administered with furosemide in comparison to naproxen and placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, non smoker male subjects aged 18 and 35 years (inclusive), at the Screening visit.
2. Body Mass Index (BMI) strictly between 18 and 30 kg/m² (inclusive) with body weight≥ 50 kg at the Screening visit.
3. Normal physical examination at the Screening visit.
4. Normal ECG (12-lead) at the Screening visit, as judged by the Investigator.
5. At Screening and run-in period visits , Systolic Blood Pressure (SBP) between 100 and 139 mmHg (inclusive) and Diastolic Blood Pressure (DBP) between 50 and 89 mmHg (inclusive).
6. At Screening and run-in period visits, HR between 45 and 90 bpm (inclusive).
7. Subjects must be able to understand the written information sheet and informed consent and comply with all study requirements.
8. Subjects must provide a written, dated and signed informed consent prior to any study procedure.

Exclusion Criteria:

1. A history of hypersensitivity reactions (such as asthma, rhinitis, or urticaria) to aspirin, naproxen or any other NSAIDs; or hypersensitivity or contraindications to organic nitrate drugs or hypersensitivity to furosemide or to sinistrine or PAH.
2. Family history of hypertension which may disqualify the subject, as judged by the investigator..
3. History of any clinically relevant gastrointestinal (such as gastritis or gastric ulcer), respiratory, psychiatric, neurologic, kidney, liver, cardiac disease, bleeding disorder, other disease/condition or abnormal physical finding which may interfere with the study objectives. The investigator may disqualify any subject for a sound medical or psychiatric reason.
4. History or presence of ASAT >40UI/L, ALAT >40UI/L, serum bilirubin 3 times above the Upper Limit of Normal range at the Screening visit.
5. Creatinine clearance inferior/equal to 80 ml/min as calculated with the Cockcroft-Gault formula (Appendix 5 of the protocol) at the Screening visit.
6. Plasmatic potassium <3.5 mmole/L at the Screening visit.
7. Seropositivity for HBs, HBc, HIV 1 or HIV 2 at the Screening visit.
8. Donations of blood, plasma or platelets within 3 months prior to the Screening visit or donation planned during the 3 months following Day 8.
9. Any clinically significant abnormal laboratory values at the Screening visit.
10. At the Screening visit, after 1 minute in a standing position, a drop of more than 20 mmHg in SBP or 10 mmHg in DBP or a clinical manifestation of postural hypotension.
11. Chronic use of any drugs (prescription or OTC) within 4 weeks prior to Visit 2 (single use of medication such as paracetamol for headache will be tolerated at the lowest possible dose).
12. Intake of any Nitric Oxide Synthase Inhibitor within 1 month before Screening visit.
13. History of drug addiction or alcohol abuse as defined by DSM IVR, diagnostic criteria for drug and alcohol abuse or drug addiction.
14. Positive drug screening (opiates, cannabinoids, cocaine, benzodiazepines, amphetamines, barbiturates) at the Screening visit.
15. Current participation or participation within 60 days prior to the Screening visit, in another investigational study, including the present study or any previous enrolment in a naproxcinod study.
16. In custody due to an administrative or a legal decision, or under tutelage, or being admitted to a sanitary or social institution.
17. Any direct or indirect involvement with the study conduct or staff at site or any family link with study site staff.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2009-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of naproxcinod on the renal function when co-administered with furosemide in comparison to naproxen and placebo | Day 8, between H3 and H9

SECONDARY OUTCOMES:
to assess the effect of naproxcinod on blood pressure (BP) in comparison with naproxen and placebo over 1 week and when co-administered with furosemide + to assess the general safety and tolerability | for over 1 week
To evaluate the effect of naproxcinod when administered alone on renal function, after a week of administration, in comparison with naproxen and placebo. | Day 8 at H4